CLINICAL TRIAL: NCT07066241
Title: Hospital, Interventional Radiology Unit
Brief Title: Virtual Reality on Stress, Pain Levels in Patients With Hyperthyroidism Undergoing Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Yavuz Uren, Principal Investigator (Dr.), Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VR - Hyperthyroidi
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Virtual Reality; Hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): During the biopsy, a video with images and sounds of nature will be shown through virtual reality glasses.
  Interventions: Device: Virtual Reality Glasses
- Control group (No Intervention): No application will be made during the biopsy procedure.

INTERVENTIONS:
Device: Virtual Reality Glasses — The Effect of Virtual Reality on Stress, Pain Levels and Vital Signs in Patients with Hyperthyroidism Undergoing Fine Needle Biopsy
  Arms: Experimental group

SUMMARY:
This study aims to investigate the effects of virtual reality on stress, pain levels and vital signs in patients diagnosed with hyperthyroidism who underwent fine needle biopsy.

DETAILED DESCRIPTION:
The specific effects of virtual reality on stress, pain levels, and vital signs during fine needle biopsy in patients with hyperthyroidism have not yet been adequately studied. This study aims to investigate the effects of virtual reality on stress, pain levels and vital signs in patients diagnosed with hyperthyroidism who underwent fine needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-80 years old
2. Agreeing to participate in the study
3. No obstacle to wearing virtual reality glasses
4. Patients undergoing biopsy for diagnostic purposes
5. No problems with vision or hearing

Exclusion Criteria:

1. Those with major psychiatric disorders
2. Those with any obstacle to communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Stress; Pain Levels | pre-intervention, post-intervention (30 mimute)
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ali Eren, Principal Investigator — yavuzuren@hotmail.com
Locations (1):
- Dursun Odabas Medical Center, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No